CLINICAL TRIAL: NCT04418739
Title: Intravenous Human Albumin In Improving Pancreaticoduodenectomy Outcomes
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: JEP-2019-796
Record Dates: First submitted 2020-03-25; First posted 2020-06-05 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Pancreaticoduodenectomy; Pancreatic Fistula; Delayed Gastric Emptying; Pancreatic Cancer; Anastomotic Leak
Keywords: Pancreaticoduodenectomy; Postoperative Pancreatic Fistula; Pancreatic Cancer; Intravenous Human Albumin
MeSH Terms: conditions — Pancreatic Fistula; Gastroparesis; Pancreatic Neoplasms; Anastomotic Leak | interventions — Serum Albumin, Human

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial conducted at the University Kebangsaan Malaysia Medical Center (UKMMC) with two arms; a control a treatment arm. The treatment arm will receive intravenous human albumin intraoperatively whilst the control arm will receive standard intraoperative fluid regimes.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (No Intervention): Standard intraoperative fluid regime
- Treatment Arm (Experimental): Intravenous human albumin 1g/kg at skin incision running at 100ml/hour
  Interventions: Drug: Human albumin

INTERVENTIONS:
Drug: Human albumin — Intravenous human albumin given at a maximum dose of 1g/kg at skin incision which is infused at 100ml/hour
  Arms: Treatment Arm

SUMMARY:
Pancreaticoduodenectomy (PD), more commonly known as Whipple's surgery is the mainstay treatment for pancreatic head and periampullary cancer. Factors contributing to PD outcomes are broadly categorized to disease-related, patient-related and operative factors. Whereas an inexhaustible list of study exists on looking at reducing PD complication rates with respect to the above-mentioned factors, it was only recently that more attention has been given to the impact of perioperative and intraoperative fluid regimes on PD outcomes. This study takes interest in the impact of intraoperative fluid regimes on PD outcomes. The objective of this investigation is to compare the outcomes with the use of intraoperative intravenous human albumin versus standard intraoperative fluid regimes.

DETAILED DESCRIPTION:
This is a randomized controlled trial being conducted at the Universiti Kebangsaan Malaysia Medical Center (UKMMC) with two arms; the control and treatment arms. The treatment arm will receive intravenous human albumin intraoperatively whilst the control arm will receive standard intraoperative fluid regimes. Primary endpoint will be overall complication rates whilst secondary endpoints are length of hospitalization, length of ICU care, duration of gastroparesis, pancreatic fistula rates, surgical site infection rates, duration of surgery and intraoperative bleeding.

Beyond the intraoperative fluid regimes, postoperative care follows the standardised UKMMC Enhanced Recovery After Surgery (ERAS) protocols which saw an improvement in overall outcomes in patients who underwent pancreaticoduodenectomies (PD). Preoperative care will include nutrition optimisation, counselling, antimicrobial prophylaxis, perioperative glycemic control and near-zero fluid balance.

Data collection will include:

i. preoperative data: age, sex, ethnicity, BMI on admission, date of admission, comorbidities and the New York Heart Association (NYHA) functional status classification. Further information will include biochemical markers such as serum albumin albumin, white cell count (WCC), renal functions.

ii. Intraoperative information: duration of surgery, estimated blood loss, pancreatic duct size, pancreatic texture, amount and type of fluid administered, fluid balances and type of anastomoses.

iii. postoperative data: fluid balances and renal function of postoperative day 1 to 3, duration of ICU stay, readmission to ICU, length of hospital stay, duration to standard feeds, grading of pancreatic fistula (where relevant), surgical site infection, duration to removal of urinary catheter, cardiac complications, renal and pulmonary complications, deep vein thrombosis, re-operation, and mortality.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing pancreaticoduodenectomy that can consent to the study

Exclusion Criteria:

* Patients with known allergy to human albumin
* Patients of American Society of Anaesthesiologist (ASA) physical status class 3 and above.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2020-01-27 (Actual); Primary Completion 2022-11-26 (Estimated); Study Completion 2022-11-26 (Estimated)

PRIMARY OUTCOMES:
Overall Complications | Postoperative complications are recorded from date of surgery to date of documented complications including death, assessed from date of surgery to date of discharge or death, whichever came earlier, for up to 12 months.
  Complications are defined as any deviation from the normal postoperative course, graded from I to V following the Clavien-Dindo classification of complications whereby Grade I are mild complications not needing any additional interventions and Grade V equates to the most severe complication which is death.

SECONDARY OUTCOMES:
Length of Hospital Stay | From date of surgery to date of discharge or date of death, whichever came earlier, assessed up to 12 months
  Duration of days of hospitalization
Length of ICU stay | From date of surgery to date of discharge or date of death, whichever came earlier, assessed up to 12 months
  Duration of stay in ICU (in days), where relevant
Postoperative Pancreatic Fistula (POPF) rates | From date of surgery to date of discharge or date of death, whichever came earlier, assessed up to 12 months
  Rates of postoperative pancreatic fistula
Delayed Gastric Emptying | From date of surgery to date of discharge or date of death, whichever came earlier, assessed up to 12 months
  Rates of prolonged gastroparesis
Ease of surgery | Duration is measured from the start time till the end time of surgery and will be assessed at the end of surgery for up to 12 months
  Measured in duration of surgery (in hours & mins)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Chik, Study Chair — Universiti Kebangsaan Malaysia Medical Center
Locations (1):
- Universiti Kebangsaan Malaysia Medical Center, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brandstrup B, Tonnesen H, Beier-Holgersen R, Hjortso E, Ording H, Lindorff-Larsen K, Rasmussen MS, Lanng C, Wallin L, Iversen LH, Gramkow CS, Okholm M, Blemmer T, Svendsen PE, Rottensten HH, Thage B, Riis J, Jeppesen IS, Teilum D, Christensen AM, Graungaard B, Pott F; Danish Study Group on Perioperative Fluid Therapy. Effects of intravenous fluid restriction on postoperative complications: comparison of two perioperative fluid regimens: a randomized assessor-blinded multicenter trial. Ann Surg. 2003 Nov;238(5):641-8. doi: 10.1097/01.sla.0000094387.50865.23. PMID 14578723
- [Result] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Result] Lassen K, Coolsen MM, Slim K, Carli F, de Aguilar-Nascimento JE, Schafer M, Parks RW, Fearon KC, Lobo DN, Demartines N, Braga M, Ljungqvist O, Dejong CH; ERAS(R) Society; European Society for Clinical Nutrition and Metabolism; International Association for Surgical Metabolism and Nutrition. Guidelines for perioperative care for pancreaticoduodenectomy: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Clin Nutr. 2012 Dec;31(6):817-30. doi: 10.1016/j.clnu.2012.08.011. Epub 2012 Sep 26. PMID 23079762
- [Result] Lavu H, Sell NM, Carter TI, Winter JM, Maguire DP, Gratch DM, Berman RA, Feil MG, Grunwald Z, Leiby BE, Pequignot EC, Rosato EL, Yeo CJ. The HYSLAR trial: a prospective randomized controlled trial of the use of a restrictive fluid regimen with 3% hypertonic saline versus lactated Ringers in patients undergoing pancreaticoduodenectomy. Ann Surg. 2014 Sep;260(3):445-53; discussion 453-5. doi: 10.1097/SLA.0000000000000872. PMID 25115420
- [Result] Boldt J. Use of albumin: an update. Br J Anaesth. 2010 Mar;104(3):276-84. doi: 10.1093/bja/aep393. Epub 2010 Jan 24. PMID 20100698 (Retraction: PMID 32861413 Br J Anaesth. 2020 Sep;125(3):417)
- [Result] Ring J, Messmer K. Incidence and severity of anaphylactoid reactions to colloid volume substitutes. Lancet. 1977 Feb 26;1(8009):466-9. doi: 10.1016/s0140-6736(77)91953-5. PMID 65572
- [Result] Ling, Q. Y., Ariffin, A. C., Azman, A., Zuhdi, Z., Othman, H., & Jarmin, R. (2017). Early postoperative outcomes for pancreaticoduodenectomy before and after implementation of enhanced recovery after surgery (ERAS) protocol. Surgical Chronicles, 22(3), 109-113
- [Result] Soar J, Pumphrey R, Cant A, Clarke S, Corbett A, Dawson P, Ewan P, Foex B, Gabbott D, Griffiths M, Hall J, Harper N, Jewkes F, Maconochie I, Mitchell S, Nasser S, Nolan J, Rylance G, Sheikh A, Unsworth DJ, Warrell D; Working Group of the Resuscitation Council (UK). Emergency treatment of anaphylactic reactions--guidelines for healthcare providers. Resuscitation. 2008 May;77(2):157-69. doi: 10.1016/j.resuscitation.2008.02.001. Epub 2008 Mar 20. PMID 18358585
- [Result] Bassi C, Marchegiani G, Dervenis C, Sarr M, Abu Hilal M, Adham M, Allen P, Andersson R, Asbun HJ, Besselink MG, Conlon K, Del Chiaro M, Falconi M, Fernandez-Cruz L, Fernandez-Del Castillo C, Fingerhut A, Friess H, Gouma DJ, Hackert T, Izbicki J, Lillemoe KD, Neoptolemos JP, Olah A, Schulick R, Shrikhande SV, Takada T, Takaori K, Traverso W, Vollmer CM, Wolfgang CL, Yeo CJ, Salvia R, Buchler M; International Study Group on Pancreatic Surgery (ISGPS). The 2016 update of the International Study Group (ISGPS) definition and grading of postoperative pancreatic fistula: 11 Years After. Surgery. 2017 Mar;161(3):584-591. doi: 10.1016/j.surg.2016.11.014. Epub 2016 Dec 28. PMID 28040257
- [Result] Wente MN, Bassi C, Dervenis C, Fingerhut A, Gouma DJ, Izbicki JR, Neoptolemos JP, Padbury RT, Sarr MG, Traverso LW, Yeo CJ, Buchler MW. Delayed gastric emptying (DGE) after pancreatic surgery: a suggested definition by the International Study Group of Pancreatic Surgery (ISGPS). Surgery. 2007 Nov;142(5):761-8. doi: 10.1016/j.surg.2007.05.005. PMID 17981197
- [Result] Laxenaire MC, Charpentier C, Feldman L. [Anaphylactoid reactions to colloid plasma substitutes: incidence, risk factors, mechanisms. A French multicenter prospective study]. Ann Fr Anesth Reanim. 1994;13(3):301-10. doi: 10.1016/s0750-7658(94)80038-3. French. PMID 7992937
- [Result] Fischer M, Matsuo K, Gonen M, Grant F, Dematteo RP, D'Angelica MI, Mascarenhas J, Brennan MF, Allen PJ, Blumgart LH, Jarnagin WR. Relationship between intraoperative fluid administration and perioperative outcome after pancreaticoduodenectomy: results of a prospective randomized trial of acute normovolemic hemodilution compared with standard intraoperative management. Ann Surg. 2010 Dec;252(6):952-8. doi: 10.1097/SLA.0b013e3181ff36b1. PMID 21107104